CLINICAL TRIAL: NCT00747409
Title: Randomized, Long-Term Study About the Effects of Analogue Versus Human Insulin Based Regimens (Insulin Detemir and Aspart Versus NPH- and Regular Human Insulin) on Metabolic Control and Myocardial Function in People With Type 2 Diabetes.
Brief Title: Insulin Effects on Metabolism and Cardiovascular Function in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Munich Municipal Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Prof. Dr. Petra-Maria Schumm-Draeger, Munich Municipal Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnaHum
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: postprandial glucose, diastolic function, analogue insulins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Detemir; Insulin; Insulin, Isophane; insulin, neutral

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hum (Active Comparator): use of human regular insulin and NPH insulin
  Interventions: Drug: human regular insulin and NPH insulin (Actrapid, Protaphne)
- Ana (Active Comparator): use of insulin aspart and insulin detemir
  Interventions: Drug: insulin aspart and detemir (NovoRapid, Levemir)

INTERVENTIONS:
Drug: insulin aspart and detemir (NovoRapid, Levemir) — use of basal-bolus therapy with insulin aspart and detemir
  Other Names: Insulin NovoRapid, Insulin Levemir
  Arms: Ana
Drug: human regular insulin and NPH insulin (Actrapid, Protaphne) — basal-bolus therapy with human regular and NPH insulin
  Other Names: Insulin Actrapid, Insulin Protaphne
  Arms: Hum

SUMMARY:
Compared to human insulins analogue insulins offer the option of optimizing metabolism also in type 2 diabetes. Especially, fast acting insulin analogues lower postprandial glucose levels more effectively than human regular insulin. However, it is not known whether therapy with analogue insulins can also improve the subclinically impaired myocardial function in type 2 diabetes. This prospective, randomized, open long term study compared the effects of a basal-bolus insulin therapy with analogue insulins versus human insulins on metabolic control and systolic and diastolic myocardial function, testing the hypothesis that optimized postprandial glucose control improves cardiac function and cardiovascular risk.

DETAILED DESCRIPTION:
This is a single centre, long term (24-48 months), therapy controlled and randomised study with blinded analysis of the ultrasound data in 120 patients with type 2 diabetes mellitus and with previous insulin therapy. After recruitment and informed consent, patients are randomized to two treatment arms according to a randomisation protocol which takes into account age and absence or presence of cardiovascular events in each patient's history.

In one treatment arm, the intensive insulin therapy is based on human insulin (insulin NPH and regular human insulin) while in the other arm, the intensive insulin therapy is based on analogue insulin (insulin detemir and insulin aspart). Both treatment arms will be titrated to identical glycemic goals (fasting blood glucose <110 mg/dL and post prandial blood glucose <150 mg/dL).

All patients will be updated in their skills of self medication by the departmental diabetic teaching programme und will receive life style instructions during each visit. Furthermore, they are encouraged to keep records of any episode of hypoglycemia throughout the study. Outpatient visits for metabolic control are every 3 months and ultrasound and blood tests every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes, insulin therapy

Exclusion Criteria:

* type 1 diabetes, BMI >40, pregnancy,

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-07; Primary Completion 2009-03 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
postprandial blood glucose at the end of the study and its change from baseline. | 24-48 months treatment period

SECONDARY OUTCOMES:
diastolic myocardial function | 24-48 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Petra-Maria Schumm-Draeger, MD, PHD, Principal Investigator — Munich Academic Teaching Hospital Bogenhausen; Helene von Bibra, MD, PHD, Study Chair — Munich Academic Teaching Hospital Bogenhausen
Locations (1):
- Staedt. Klinikum Muenchen Bogenhausen, Munich, Bavaria, Germany

REFERENCES:
- [Background] Bretzel RG, Arnolds S, Medding J, Linn T. A direct efficacy and safety comparison of insulin aspart, human soluble insulin, and human premix insulin (70/30) in patients with type 2 diabetes. Diabetes Care. 2004 May;27(5):1023-7. doi: 10.2337/diacare.27.5.1023. PMID 15111514
- [Background] von Bibra H, Hansen A, Dounis V, Bystedt T, Malmberg K, Ryden L. Augmented metabolic control improves myocardial diastolic function and perfusion in patients with non-insulin dependent diabetes. Heart. 2004 Dec;90(12):1483-4. doi: 10.1136/hrt.2003.020842. No abstract available. PMID 15547039
- [Background] Shaw JE, Hodge AM, de Courten M, Chitson P, Zimmet PZ. Isolated post-challenge hyperglycaemia confirmed as a risk factor for mortality. Diabetologia. 1999 Sep;42(9):1050-4. doi: 10.1007/s001250051269. PMID 10447514
- [Derived] von Bibra H, Siegmund T, Kingreen I, Riemer M, Schuster T, Schumm-Draeger PM. Effects of analogue insulin in multiple daily injection therapy of type 2 diabetes on postprandial glucose control and cardiac function compared to human insulin: a randomized controlled long-term study. Cardiovasc Diabetol. 2016 Jan 16;15:7. doi: 10.1186/s12933-015-0320-2. PMID 26772807